CLINICAL TRIAL: NCT02177071
Title: A proSpective Randomized Controlled Trial comParing infliximAb-antimetabolites Combination Therapy to Anti-metabolites monotheRapy and Infliximab monothErapy in Crohn's Disease Patients in Sustained Steroid-free Remission on Combination Therapy
Acronym: SPARE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Collaborators: Saint-Louis Hospital, Paris, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GETAID 2014-03
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Crohn's Disease
Keywords: CROHN DISEASE; INFLIXIMAB; COMBINATION THERAPY; steroid free remission; anti-metabolites
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab; Azathioprine; Mercaptopurine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- INFLIXIMAB AND ANTI METABOLITE (No Intervention): continuing scheduled infliximab treatment and anti-metabolite
- STOP INFLIXIMAB CONTINUING ANTI METABOLITE (Other): discontinuing infliximab and continuing the anti-metabolite
  Interventions: Drug: INFLIXIMAB
- CONTINUING INFLIXIMAB AND discontinuing anti-metabolites (Other): CONTINUING INFLIXIMAB AND DISCONTINUING ANTI METABOLITE
  Interventions: Drug: AZATHIOPRINE; Drug: MERCAPTOPURINE; Drug: Methotrexate

INTERVENTIONS:
Drug: INFLIXIMAB
  Arms: STOP INFLIXIMAB CONTINUING ANTI METABOLITE
Drug: AZATHIOPRINE
  Arms: CONTINUING INFLIXIMAB AND discontinuing anti-metabolites
Drug: MERCAPTOPURINE
  Arms: CONTINUING INFLIXIMAB AND discontinuing anti-metabolites
Drug: Methotrexate
  Arms: CONTINUING INFLIXIMAB AND discontinuing anti-metabolites

SUMMARY:
Phase IV

Design : Prospective, open-label, randomized three-arms study

Main Inclusion criteria Luminal Crohn's disease patients with steroid free remission for at least 6 months and a combination therapy with infliximab and anti-metabolites for at least 8 months

Primary objective To demonstrate that Infliximab scheduled maintenance with or without antimetabolites is superior to antimetabolites alone to maintain sustained steroid-free remission over 2 years, while the latter is non inferior with regards to the mean time spent in remission over the same duration

Main co-primary end points Clinical relapse rate at 2 years Mean remission duration within 2 years Study treatment Infliximab, Mercaptopurine, azathioprine, methotrexate.

Number of subjects 225 randomized patients (75 per arm)

Study duration: 3 + 2 years Enrollment: 3 years Follow-up: 2 years

DETAILED DESCRIPTION:
3. STUDY OBJECTIVES 3.1. Primary objective To assess the effect of two withdrawal strategies over two years in patients with stable remission for more than 6 months on combination therapy with infliximab and antimetabolites, and demonstrate that continued combination of infliximab and antimetabolites or continued monotherapy with infliximab are both superior to antimetabolites alone for maintaining sustained steroid-free clinical remission, while antimetabolites alone are non-inferior with regards to the mean time spent in remission 3.2. Secondary objectives

* To identify baseline predictive factors of relapse in the three study groups.
* To assess the ability of blood CRP and fecal calprotectin to predict short term relapse in the three groups.
* To assess time spent inclinical remission in the three groups.
* To assess the rate of treatment failure in the three study groups.
* To assess the time to treatment failure in the three study groups.
* To assess progression of bowel damage in the three groups.
* To assess the safety and efficacy of infliximab retreatment in the antimetabolites group.
* To assess safety in the three study groups.
* To assess the health related quality of life in the three study groups.
* To assess direct and indirect costs in the three study groups.
* To assess evolution of blood CRP and fecal calprotectin in the three study groups.
* To assess evolution of infliximab trough levels and ATI in the two infliximab scheduled maintenance groups.
* To assess genetic association with the various clinical and biological outcomes.
* To assess the impact of 6TGN levels on the various clinical and biological outcomes in the purine treated patients 4. STUDY POPULATION 4.1. Selection of study population Patients to be included are those who have been in steroid free remission for at least 6 months and with scheduled infliximab/antimetabolites combination therapy for at least 8 months, with a scheduled infliximab treatment administrated every 8 weeks for the last 4 months.

4.2. Source of recruitment Patients are recruited from participating GETAID IBD-centers in France, Belgium and SOIBD IBD-centers in Sweden, and selected centres in UK, Germany, Netherland and Australia 4.3. Inclusion criteria

To be eligible all of the following criteria must be met:

* Diagnosis of Crohn's disease.
* Male or female, age > 18 years.
* Currently treated with a combination therapy with infliximab and anti-metabolites for luminal Crohn's disease.
* Combined therapy with scheduled infliximab and anti-metabolites for at least 8 months.
* Scheduled administration of infliximab 5 mg/Kg every 8 weeks over the last 4 months.
* Antimetabolites administered at a stable dosage for the last 3 months: at least 1 mg/Kg or 2 mg/Kg for mercaptopurine and azathioprine, respectively, or the highest tolerated dosage if intolerance to standard dose;(lower dose than standard dose is also allowed if 6 TGN > 235 pmol) ; at least 15 mg/week subcutaneously for methotrexate.
* Patients in steroid free clinical remission for at least 6 months according to retrospective assessment of the patients' files.
* CDAI < 150 at baseline.
* A contraceptive during the whole study
* Patients able to understand the information provided to them and to give written informed consent for the study

4.4. Exclusion criteria

* Patients who have presented a severe acute or delayed reaction to infliximab.
* Perianal fistulae as the main indication for infliximab treatment
* Active perianal/abdominal fistulae at time of inclusion, defined by active drainage
* Patients with ostomy or ileoanal pouch
* Pregnancy or planned pregnancy during the study
* Inability to follow study procedures as judged by the investigator
* Non-compliant subjects.
* Participation in another therapeutic study

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn's disease.
* Male or female, age > 18 years.
* Currently treated with a combination therapy with infliximab and anti-metabolites for luminal Crohn's disease.
* Combined therapy with scheduled infliximab and anti-metabolites for at least 8 months.
* Scheduled administration of infliximab 5 mg/Kg every 8 weeks over the last 4 months.
* Antimetabolites administered at a stable dosage for the last 3 months: at least 1 mg/Kg or 2 mg/Kg for mercaptopurine and azathioprine, respectively, or the highest tolerated dosage if intolerance to standard dose; at least 15 mg/week subcutaneously for methotrexate.
* Patients in steroid free clinical remission for at least 6 months according to retrospective assessment of the patients' files.
* CDAI < 150 at baseline.
* A contraceptive during the whole study for childbearing potential female patients.
* Patients able to understand the information provided to them and to give written informed consent for the study

Exclusion Criteria:

* Patients who have presented a severe acute or delayed reaction to infliximab.
* Perianal fistulae as the main indication for infliximab treatment
* Active perianal/abdominal fistulae at time of inclusion, defined by active drainage
* Patients with ostomy or ileoanal pouch
* Pregnancy or planned pregnancy during the study
* Inability to follow study procedures as judged by the investigator
* Non-compliant subjects.
* Participation in another therapeutic study
* Steroid use ≤6 months prior to screening
* Currently receiving steroids, immunosuppressive agents (other than purine, methotrexate), biologic treatment (other than infliximab) or thalidomide

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2015-10-09 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
co-primary efficacy end points | 2 ans
  There will be two co-primary efficacy end points
  Relapse rate at 2 years, relapse being defined by either one of the following events:
  * A CDAI>250 at any visit or between 150 and 250 with an increase of at least 70 points, over two consecutive visits one week apart associated with a CRP > 5 mg/l or a fecal calprotectin > 250 microg/g
  * A new opening fistula, perianal or entero-cutaneous.
  * An intra-abdominal abcess (size of at least 3 cm) or perianal abcess (size of at least 2 cm)
  * An episode of intestinal obstruction due to Crohn's lesions confirmed by medical imaging and requiring hospitalisation (also considered as treatment failure, see below)
  Mean restricted time spent in remission This time will be computed in all patients, from baseline (CDAI <150 and with absence of fistula drainage) until relapse, as defined above, within the 2 first years. First and subsequent remissions will be summed up within the two first years.

SECONDARY OUTCOMES:
relapse in each arm. | 2 years
  * Time to relapse in each arm.
  * Factors associated with time to relapse.
  * Time to relapse according to CRP and calprotectin value measured every 2 months over the follow up.
Sustained clinical remission | 2years
  Sustained clinical remission defined by CDAI<150 without steroids over two years.
Treatment failure | 2 years
  * Treatment failure rate. Treatment failure is defined by not achieving remission after treatment adaptation following a relapse according to protocol (CDAI<150 or, in case of relapse defined by the occurence of a new fistula, the absence of fistula closure). The occurence of an intra-abdominal or peri-anal abcess and the occurence of an intestinal obstruction due to Crohn's lesions and requiring a surgical resection or an endoscopic dilatation are also directly considered as treatment failure and will not be managed by treatment adaptation according to protocol.
  * Time to treatment failure.
Tissue damage progression | 2 years
  - Tissue damage progression will be assessed by the Lémann Score absolute and relative change between baseline and en of the study (2 years).
Endoscopic remission | 2 years
  Endoscopic remission at the end of study

OTHER OUTCOMES:
disability index | 2 YEARS
  disability index
adverse events and SAE | 2 YEARS
  adverse events and SAE, events related to re-infusions,
BIOLOGICS | 2 YEARS
  trough levels of infliximab, ATI , hsCRP, fecal calprotectin
SCORES AND COST | 2 YEARS
  direct medical costs, work productivity and activity index, short IBDQ

CONTACTS AND LOCATIONS:
Overall Officials: David Laharie, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives
Locations (27):
- St Vincent Hospital, Melbourne, Australia
- Belgium (2):
  - CHU LIEGE - Sart Tilman, Liège, Province De Liège
  - Gent University Hospital, Ghent
- France (24):
  - Chu Clermont-Ferrand, Clermont-Ferrand, Auvergne-Rhône-Alpes
  - CHU LYON, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Chu Saint Etienne, Saint-Etienne, Auvergne-Rhône-Alpes
  - Chu Besancon, Besançon, Bourgogne-Franche-Comté
  - Chu Rennes, Rennes, Brittany Region
  - Chu Tours, Tours, Centre-Val de Loire
  - Chu Reims, Reims, Grand Est
  - Chu Nancy, Vandœuvre-lès-Nancy, Grand Est
  - Chu Amiens, Amiens, Hauts-de-France
  - Chu Lille, Lille, Hauts-de-France
  - Chr Valencienne, Valenciennes, Hauts-de-France
  - Caen Unversity Hospital, Caen, Normandy
  - CHU Bordeaux - Pessac, Pessac, Nouvelle-Aquitaine
  - Chu Montpellier, Montpellier, Occitanie
  - Chu Toulouse, Toulouse, Occitanie
  - Chu Nantes, Nantes, Pays de la Loire Region
  - CHU NICE, Nice, Provences Alpes Cote d'Azur
  - Hopital Saint Joseph, Paris
  - Hopital Beaujon, Clichy, Île-de-France Region
  - Chu Kremlin Bicetre, Le Kremlin-Bicêtre, Île-de-France Region
  - Hopital Bicetre, Le Kremlin-Bicêtre, Île-de-France Region
  - Hopital Saint Louis, Paris, Île-de-France Region
  - Hopital St Antoine, Paris, Île-de-France Region
  - Montsouris Mutualist Institute, Paris, Île-de-France Region

REFERENCES:
- [Derived] Pierre N, Huynh-Thu VA, Baiwir D, Mazzucchelli G, Fleron M, Trzpiot L, Eppe G, De Pauw E, Laharie D, Satsangi J, Bossuyt P, Vuitton L, Vieujean S, Colombel JF, Meuwis MA, Louis E; GETAID and the SPARE-Biocycle research group. External validation of serum biomarkers predicting short-term and mid/long-term relapse in patients with Crohn's disease stopping infliximab. Gut. 2024 Nov 11;73(12):1965-1973. doi: 10.1136/gutjnl-2024-332648. PMID 39134391
- [Derived] Louis E, Resche-Rigon M, Laharie D, Satsangi J, Ding N, Siegmund B, D'Haens G, Picon L, Bossuyt P, Vuitton L, Irving P, Viennot S, Lamb CA, Pollok R, Baert F, Nachury M, Fumery M, Gilletta C, Almer S, Ben-Horin S, Bouhnik Y, Colombel JF, Hertervig E; GETAID and the SPARE-Biocycle research group. Withdrawal of infliximab or concomitant immunosuppressant therapy in patients with Crohn's disease on combination therapy (SPARE): a multicentre, open-label, randomised controlled trial. Lancet Gastroenterol Hepatol. 2023 Mar;8(3):215-227. doi: 10.1016/S2468-1253(22)00385-5. Epub 2023 Jan 11. PMID 36640794
- [Derived] Hirten RP, Lakatos PL, Halfvarson J, Colombel JF. Reply. Clin Gastroenterol Hepatol. 2021 Jun;19(6):1301-1302. doi: 10.1016/j.cgh.2020.07.061. Epub 2020 Nov 26. No abstract available. PMID 33248096